CLINICAL TRIAL: NCT03882528
Title: Bridging Trial to Evaluate the Infectivity Equivalence of Current and New Lots of Plasmodium Falciparum Strain NF54 (Clone 3D7) Within the WRAIR Controlled Human Malaria Infection (CHMI) Model
Brief Title: Evaluate the Infectivity Equivalence of Current and New Lots of Plasmodium Falciparum Strain NF54
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: S-18-02
Record Dates: First submitted 2018-10-24; First posted 2019-03-20 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Infective controls (Experimental): Controlled Human Malaria Infection (CHMI) will consist of exposure to Plasmodium falciparum sporozoites through the bites of infected mosquitoes. Beginning 5 days after the challenge, subjects will be evaluated daily for the development of malaria infection using a blood smear.
  Interventions: Biological: Plasmodium falciparum malaria parasite

INTERVENTIONS:
Biological: Plasmodium falciparum malaria parasite — Laboratory cultured Plasmodium falciparum strain 3D7 delivered via the bite of 5 infected mosquitoes with salivary gland scores of at least 2+ (11-100 sporozoites observed).

SUMMARY:
Objectives:

Primary:

• To characterize the infectivity of the new lot of Plasmodium falciparum strain 3D7 within the standard WRAIR CHMI model as compared to the current lot (historical data)

Secondary:

* To assess safety of the new lot of P falciparum parasites
* To assess the kinetics of detecting parasitemia and parasite clearance by quantitative polymerase chain reaction (qPCR) as compared to blood smear
* To obtain plasma samples to restore the testing control pool for malaria serology testing and for future malaria research

DETAILED DESCRIPTION:
This is a single center, open label CHMI study. CHMI will consist of exposure to Plasmodium falciparum sporozoites through the bites of infected mosquitoes. After the challenge, subjects will be evaluated daily for the development of malaria infection using a blood smear. Unless previously diagnosed and fully treated, subjects will be required to stay in a hotel for a maximum of 12 nights starting on or around the evening of Day 7 post challenge.

All subjects diagnosed with malaria infection based on smears will be prescribed a standard malaria treatment regimen to begin on the day that parasitemia is detected. Subjects who do not become parasitemic (via smear) by Day 19 will be empirically treated for malaria.

After the hotel phase, all challenged subjects will have a final scheduled follow-up visit on Day 28 (±7 days).

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, you must meet ALL of the following conditions:

  * You are between the ages of 18 and 50 years old.
  * You are willing and able to participate in all planned study visits for the duration of the study.
  * You are in good general health based on your medical history, physical examination, EKG, and screening laboratories.
  * You are able to understand and sign this informed consent.
  * You pass the written test called the 'Assessment of Understanding' with a score of at least 80% (8 out of 10 questions correct).
  * You agree not to donate blood during the study and for 3 years after the malaria challenge.
  * You agree not to travel to place(s) where there is malaria during the time of the study.
  * If you are a female, you must agree to consistently use effective birth control (e.g., oral or implanted contraceptives, intrauterine device (IUD), diaphragm with spermicide, abstinence, cervical cap) during the period from the day of screening (today) through 3 months after the malaria challenge.
  * You must be willing to take anti-malarial treatment after CHMI, if indicated.
  * You must agree to stay in a pre-determined hotel near the NMRC CTC during the designated post-CHMI follow-up period from approximately 7 days after malaria challenge until antimalarial treatment is completed, if indicated.
  * If you are an active duty military or federal employee, you must have approval from your supervisory chain to participate. The appropriate approval form will be provided to you.

Exclusion Criteria:

* You must not have any of the following:

  * Any history of malaria infection or having been given a malaria vaccine
  * Any history travel to a country with falciparum malaria in the past 6 months, or planned travel to such an area during the course of the study
  * Any history of having lived in an area with falciparum malaria for more than 5 years.
  * Any use of medications that prevent or treat malaria during the 1 month prior to challenge or planned use during the study (outside of the drugs provided by the study team).
  * Any serious medical illness or condition involving the heart, liver, lungs, or kidneys
  * Any significant risk for developing heart disease in the next 5 years. The risk for developing heart disease in the next 5 years will be determined by a combination of the following factors: high blood pressure, smoking, weight, family history of heart disease and the presence of diabetes
  * Any medical illness or condition involving your blood or immune system (to include sickle cell trait or thalassemia trait)
  * Any abnormal (as determined by a physician) screening laboratory test results
  * Any history of neurologic disease (including migraines or seizures)
  * Any history of psoriasis (itchy skin rash) or porphyria (rare disturbance of metabolism), since these conditions could get worse after treatment with chloroquine (a medication for treating malaria).
  * You have had your spleen removed
  * Any past or current infection with HIV, Hepatitis C, or Hepatitis B
  * Any use of investigational drugs or vaccines within 1 month before starting the study
  * Any allergy to or inability to take the anti-malaria medications used in this study
  * Any history of allergic reaction to mosquito bites that required hospitalization
  * You must not be pregnant or nursing, or have any plans to become pregnant or breastfeed during the period from now through 3 months after malaria challenge
  * Any chronic use of steroids or other medications that affect the immune system in the 6 months before malaria challenge. Inhaled and topical (used on the skin) steroids are allowed.
  * You plan to have surgery between enrollment and 3 months after malaria challenge.
  * Any active alcohol or drug abuse
  * You have any other physical or psychologic condition or laboratory abnormality that the study doctor thinks may increase your risk of having side effects or compromise the results of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Moon, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infective Controls
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy, malaria-naïve adults (males and non-pregnant, non-lactating females), aged 18 to 50 years old (inclusive) were recruited from the Washington/ Baltimore DC metropolitan area to participate in this Controlled Human Malaria Infection (CHMI) study. Up to 12 subjects were enrolled (defined as having undergone malaria challenge) into this trial. All 12 subjects were challenged with the new lot of female Anopheles mosquitoes infected with Plasmodium falciparum strain NF54 (clone 3D7), lot 1887
Arm/Group | Infective Controls
Number analyzed (Participants) | 12
Age, Customized [Mean (Standard Deviation); unit: years] — Healthy, malaria-naïve adults aged 18 to 50 years old
  years
    Age | 28.7 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: To Characterize the Infectivity of a New Lot of Plasmodium Falciparum Strain 3D7 Developing Parasitemia Within the Standard WRAIR CHMI Model.
Description: Number of challenged subjects exposed to the new lot of Plasmodium falciparum strain 3D7 parasites developing parasitemia (defined as 2 unambiguous malaria parasites on a single smear).
Time Frame: Within 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Infective Controls
Number analyzed (Participants) | 12
Participants
  9 Days post-challenge | 0
  10 Days post-challenge | 1
  11 Days post-challenge | 5
  12 Days post-challenge | 5
  13 Days post-challenge | 0
  14 Days post-challenge | 1

2. Secondary Outcome: Diagnostic Efficacy; Time to Parasitemia by Blood Smear Method After the P Falciparum Challenge
Description: Time to parasitemia by blood smear method after the P falciparum challenge. Time to parasitemia is defined as the time from CHMI to a first positive malaria parasite result. Parasitemia was defined as the presence of 2 unambiguous malaria parasites on a single smear. Beginning on Day 1 after their challenge, subjects were seen and evaluated daily by a study investigator and blood was drawn for determination of parasitemia by qPCR. Beginning on Day 5 and through Day 19 after their challenge, blood from these daily draws was utilized to generate blood smears to evaluate the development of malaria infection. In addition to smears, subjects were also evaluated for the presence of parasitemia via qPCR. In addition to smears, subjects were also evaluated for the presence of parasitemia via qPCR. However, only blood smears were used for diagnosis during this trial and evaluation of treatment success.
Time Frame: Within 2-3 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infective Controls
Number analyzed (Participants) | 12
days | 11.6 (1.00)

3. Secondary Outcome: Diagnostic Efficacy; Time to Parasitemia (Days) by qPCR Method After the P Falciparum Challenge
Description: Time to parasitemia by qPCR method after the P falciparum challenge. Time to parasitemia is defined as the time from CHMI to a first positive malaria parasite result. Parasitemia was defined as the presence of 2 unambiguous malaria parasites on a single smear. On Day 0, subjects were evaluated by qPCR once prior to challenge, to establish a baseline. Beginning on Day 1 through Day 19 after their challenge, subjects were seen and evaluated daily by a study investigator and blood was drawn for determination of parasitemia by qPCR. Beginning on Day 5 and going through Day 19 after their challenge, blood from these daily draws was utilized to generate blood smears to evaluate the development of malaria infection. In addition to smears, subjects were also evaluated for the presence of parasitemia via qPCR. However, only blood smears were used for diagnosis during this trial and evaluation of treatment success.
Time Frame: Within 2-3 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infective Controls
Number analyzed (Participants) | 12
days | 7.3 (0.65)

4. Secondary Outcome: Diagnostic Efficacy; Quantification of Parasite Clearance Time (PCT) by Blood Smear and qPCR Methods After Initiation of Antimalarial Treatment
Description: Time to Clearance was determined for all subjects for both smear and qPCR. Time to Clearance was defined as the time (in Days) from malaria diagnosis to confirmed clearance of parasitemia. Confirmed clearance of parasitemia by malaria smear was defined as the observation of 3 sequential negative (no parasites observed) daily smears. Confirmed clearance of parasitemia by qPCR was defined as 2 sequential daily (approximately 24 hours apart) negative qPCR assay results. For clarity, the day of the final test in each sequence (smear, PCR) was used as the day of confirmed clearance for calculation purposes.
Time Frame: Within 6 weeks
Population: Unless previously diagnosed and fully treated, subjects stayed in a hotel starting on the evening of Day 9 post challenge. Subjects diagnosed with malaria were treated on the day parasitemia was detected. Subjects not parasitemic by Day 19 were treated for malaria and released from the hotel. These subjects had clinic daily for completion of treatment and blood collection until treatment efficacy criteria were met. All challenged subjects had a final follow-up visit on Day 28 (±7 days).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infective Controls
Number analyzed (Participants) | 12
days
  Blood smear Method | 1.2 (0.39)
  qPCR method | 3.0 (0.60)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 35
Description: Subjects were seen and evaluated daily and adverse event reporting collected
Arm/Group | Infective Controls
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infective Controls (N=12)
Malaria (Infections and infestations) | 12
Administration site pruritus (General disorders) | 8
Administration site erythema (General disorders) | 1
Fatigue (General disorders) | 2
Headache (Nervous system disorders) | 4
Pyrexia (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Tachycardia (Cardiac disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Influenza (Infections and infestations) | 1
Alanine Aminotransferase Elevation (Investigations) | 1
Syncope (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT03882528/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT03882528/SAP_001.pdf
  • Informed Consent Form (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT03882528/ICF_002.pdf